CLINICAL TRIAL: NCT01266096
Title: PET Imaging of Patients With Melanoma and Malignant Brain Tumors Using an 124I-labeled cRGDY Silica Nanomolecular Particle Tracer: A Microdosing Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-155
Record Dates: First submitted 2010-12-21; First posted 2010-12-24 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Newly Diagnosed or Recurrent Metastatic Melanoma Patients; Malignant Brain Tumors
Keywords: 124I-cRGDY-PEG-dots; Pet scan; 10-155; melanoma; brain
MeSH Terms: conditions — Melanoma | interventions — Magnetic Resonance Spectroscopy

ARMS (1):
- newly diagnosed or recurrent head/neck melanoma (Experimental): This is a two-year microdosing study that will enroll 5 metastatic melanoma patients and 18 malignant brain tumor patients (surgical (n=13) and non-surgical candidates (n=5)). We have already accrued 5 melanoma patients and expect to accrue brain tumor patients within a 1 year period.
  Interventions: Drug: PET scan with 124I-cRGDY-PEG-dots

INTERVENTIONS:
Drug: PET scan with 124I-cRGDY-PEG-dots — Five (5) patients with newly diagnosed or recurrent melanoma, and 18 malignant brain tumor patients (surgical (n=13) or non-surgical candidates (n=5)). Patients with either primary or metastatic brain tumors, will be i.v. injected with approximately 5 mCi (3.4-6.7 nanomoles) of 124I-cRGDY-PEG-dots (specific activity range 750.0 - 1450 mCi/mol) and undergo the microdosing study for purposes of collecting pharmacokinetic and dosimetry data. All studies will be performed using a dedicated scanner, which integrates a dedicated PET scanner and a spiral CT with proprietary fusion software.

SUMMARY:
Current tests to detect cancer, including CAT scans and MRI scans, are limited. PET scans use special dyes that are injected into a vein and can better localize possible cancer. The investigators have developed a new particle that can carry a radioactive dye to a very specific area of the tumor. When using a PET scan the radioactive dye can be viewed in areas of possible disease. This particle has been studied in mice and was safe.

The particles will not treat the cancer and any images or information found during this study will not be used for your treatment. The information collected may be used to guide the design of future studies to detect and/or treat tumors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed diagnosis of melanoma or malignant brain tumor at MSKCC
* Newly-diagnosed or recurrent (local,regional, metastatic) metastatic melanoma or malignant brain tumor patients with
* Residual clinically or radiographically evident tumor, including primary cutaneous and mucosal melanomas or malignant brain tumor
* Prior radiation therapy, chemotherapy, or surgery in patients requiring flap reconstruction in the head and neck region.
* Newly diagnosed patients with previous excisional biopsy.
* Normal baseline cardiac function based upon pre-operative evaluation
* At the discretion of the physician ANC>1000/mcl and platelets>100,000/mcl.
* At the discretion of the physician Bilirubin level of < 2.0 mg/dl in the absence of a history of Gilbert's disease (or pattern consistent with Gilbert's).
* If patients have a history of malignancy other than melanoma or malignant brain tumor they must be disease-free (excluding primary cancer for metastatic patients) for ≥ 5 years at the time of enrollment.
* All patients of childbearing and child-creating age must be using an acceptable form of birth control
* Women who are pre-menopausal must have a negative serum pregnancy test

Exclusion Criteria:

* Abnormal thyroid function, such as untreated clinical diagnosis of hypothyroidism, hyperthyroidism, or other thyroid disease
* Known pregnancy or breast-feeding.
* Medical illness unrelated to the tumor which in the opinion of the attending physician and principal investigator will preclude administration of the tracer. This includes patients with uncontrolled infection, chronic renal insufficiency, myocardial infarction within the past 6 months, unstable angina, cardiac arrhythmias other than chronic atrial fibrillation and chronic active or persistent hepatitis, or New York Heart Association Classification III or IV heart disease.
* History of any malignancy (excluding primary cancer for metastatic patients) other than melanoma or malignant brain tumors for which the disease-free interval is <5 years.
* Allergic reaction to iodine-containing contrast material
* Weight greater than the 400-lb weight limit of the PET scanner
* Claustrophobia
* Inability to lie in the scanner for 30 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Conduct pilot single-dose studies of 124I-cRGDY-PEG-dots† | 2 years
  in a limited number of human melanoma and brain tumor patients to characterize biodistribution, pharmacokinetics, and metabolic stability.

SECONDARY OUTCOMES:
Estimate the radiation dosimetry of i.v.-injected 124I-cRGDY-PEG-dots. | 1 year
  studies have demonstrated that a dose 100 times the proposed human dose equivalent did not induce adverse effects
Assay particle tracer tissue distributions in tumor tissue specimens | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hilda Stambuk, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Phillips E, Penate-Medina O, Zanzonico PB, Carvajal RD, Mohan P, Ye Y, Humm J, Gonen M, Kalaigian H, Schoder H, Strauss HW, Larson SM, Wiesner U, Bradbury MS. Clinical translation of an ultrasmall inorganic optical-PET imaging nanoparticle probe. Sci Transl Med. 2014 Oct 29;6(260):260ra149. doi: 10.1126/scitranslmed.3009524. Epub 2014 Oct 29. PMID 25355699
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm